CLINICAL TRIAL: NCT06147219
Title: Primary Dynamization Versus Standard Interlocking Intramedullary Nail in Treatment of Tibial Shaft Fractures in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Salah Hafez, Resident of Orthopaedic department, Sohag University Hospitals, Sohag University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-010-04
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Tibial Shaft Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- primary dynamization interlocking intramedullary tibial nail (Active Comparator)
  Interventions: Procedure: interlocking intramedullary tibial nail
- standard interlocking intramedullary tibial nail (Active Comparator)
  Interventions: Procedure: interlocking intramedullary tibial nail

INTERVENTIONS:
Procedure: interlocking intramedullary tibial nail — primary dynamization versus standard interlocking intramedullary tibial nail

SUMMARY:
fracture shfat tibia in adults treated by interlocking intramedullary nail by primary dynamic versus standard ways

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18-50) fractures with mid shaft or distal shaft tibial fracture AO type A1, A2 and A3 and minimal soft tisuue damage

Exclusion Criteria:

* patients with comminuted fractures , old age more than 50 years , sclerotic bone , osteoporosis, osteopetrosis and bone deformity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary Dynamization Interlocking Intramedullary Tibial Nail | 12 months
  use only distal screws away from fracture site

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Whelan DB, Bhandari M, Stephen D, Kreder H, McKee MD, Zdero R, Schemitsch EH. Development of the radiographic union score for tibial fractures for the assessment of tibial fracture healing after intramedullary fixation. J Trauma. 2010 Mar;68(3):629-32. doi: 10.1097/TA.0b013e3181a7c16d. PMID 19996801
- [Background] Fracture and dislocation compendium. Orthopaedic Trauma Association Committee for Coding and Classification. J Orthop Trauma. 1996;10 Suppl 1:v-ix, 1-154. No abstract available. PMID 8814583
- [Background] Omerovic D, Lazovic F, Hadzimehmedagic A. Static or dynamic intramedullary nailing of femur and tibia. Med Arch. 2015 Apr;69(2):110-3. doi: 10.5455/medarh.2015.69.110-113. Epub 2015 Apr 6. PMID 26005261
- [Background] Vaughn J, Gotha H, Cohen E, Fantry AJ, Feller RJ, Van Meter J, Hayda R, Born CT. Nail Dynamization for Delayed Union and Nonunion in Femur and Tibia Fractures. Orthopedics. 2016 Nov 1;39(6):e1117-e1123. doi: 10.3928/01477447-20160819-01. Epub 2016 Aug 30. PMID 27575039
- [Derived] Elsayed M, Khalefa AH, Mazen MSH, Ahmed KFE. Primary dynamization versus standard static interlocking nailing in treatment of tibial shaft fractures in adults: a randomized controlled trial. BMC Musculoskelet Disord. 2025 Dec 12. doi: 10.1186/s12891-025-09376-3. Online ahead of print. PMID 41387845